CLINICAL TRIAL: NCT05268328
Title: The Effect of Foot Reflexology After Cesarean Section on Pain, Intestinal Motility and Comfort
Brief Title: The Effect of Foot Reflexology After Cesarean Section
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nülüfer Erbil (Other)
Responsible Party: Sponsor-Investigator, Nülüfer Erbil, Prof. Dr., Ordu University
Organization: Ordu University (Other)
Other Study IDs: eylul1
Record Dates: First submitted 2022-01-31; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Pain; Gastrointestinal Motility Disorder
Keywords: Cesarean section; Foot reflexology; Postpartum pain; Postpartum Comfort; nursing; Bowel problems
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Standardized, quality and evidence-based nursing care after cesarean section is important to prevent or minimize complications that may occur after cesarean section. This evidence-based care will contribute to the shortening of the recovery period of the mother, the early start of postpartum bowel movements, the decrease in the perceived pain level, and the increase in postpartum comfort, thus facilitating the adaptation to new life and roles. On the other hand, although a limited number of studies reported the effects of reflexology, no study investigating the effect of reflexology on pain, comfort level and GIS motility developed after SD was found. In this study, it was aimed to determine the effect of foot reflexology on pain, intestinal motility and comfort after cesarean section.

Hypothesis(s):

H1: Foot reflexology after cesarean section reduces the level of pain perception.

H2: Foot reflexology after cesarean section increases intestinal motility. H3: Foot reflexology after cesarean section increases postpartum comfort.

ELIGIBILITY:
Inclusion Criteria

* 18 and over,
* Performing SD under general anesthesia,
* Cesarean section at 37-42 weeks of gestation,
* The only live SD made,
* Written / verbal communication can be established,
* At least primary school graduate,
* Not having any problems during her pregnancy,
* Women who agree to participate in the study will be taken into the sample. Exclusion Criteria
* Being under 18 years old,
* Those who gave birth by cesarean section before 37-42 weeks of gestation,
* Having chronic constipation, diarrhea and using any laxative type medication,
* Having problems such as fractures, dislocations, arthritis, phlebitis, wounds, burns, fungus, eczema, inflammation in the foot tissue,
* Having cardiovascular system disease,

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women who have had cesarean section
Study Population: women who have had cesarean section
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum Comfort Scale | 3 hour
  t consists of 34 items. A 5-point Likert-type scale scoring system was used, which will enable an evaluation to be made for each item that determines the situation to be measured. For each item, expression and scoring ranging from "strongly agree" (5 points) to "strongly disagree" (1 point) were made. I totally agree with positive sentences shows the best comfort (5 points), and negative sentences show low comfort (1 point). Accordingly, the lowest score to be taken from the scale is 34, and the highest score is 170. The average value is determined by dividing the total score obtained from the scale by the number of items, and the result is shown in the 1-5 distribution. Basically, low comfort is expressed by 1 and high comfort by 5. Since the scale is gathered under three factors, it can evaluate postpartum comfort in 3 dimensions (physical, psychospiritual, sociocultural).
Visual Analog Scale | 3 hour
  Visual Analog Scale A ruler that is 10 cm or 100 mm long, with painlessness (0, zero) on one end and the highest possible pain (10, ten) on the other end, can be used horizontally or vertically. It is stated that vertical use of the scale is more appropriate because it gives quick results and is easy to apply. In this study, the vertical form of the scale will be used. Clina et al. (1992) evaluated the VAS results as 0 cm "no pain", 0.5-3 cm "mild pain", 3.5-6.5 cm "moderate pain", 7-10 cm "severe pain". A new VAS form will be used in each application so that the woman can see her previous pain score and not be affected by it.
Bowel Movements Monitoring Form | 3 hour
  the time when women's bowel movements begin to be heard, when gas is removed, and when bowel emptying occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Nülüfer Erbil, Prof. Dr., Principal Investigator — Ordu University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Altraigey A, Ellaithy M, Atia H, Abdelrehim W, Abbas AM, Asiri M. The effect of gum chewing on the return of bowel motility after planned cesarean delivery: a randomized controlled trial. J Matern Fetal Neonatal Med. 2020 May;33(10):1670-1677. doi: 10.1080/14767058.2018.1526913. Epub 2018 Oct 29. PMID 30231787
- [Result] Dikmen HA, Terzioglu F. Effects of Reflexology and Progressive Muscle Relaxation on Pain, Fatigue, and Quality of Life during Chemotherapy in Gynecologic Cancer Patients. Pain Manag Nurs. 2019 Feb;20(1):47-53. doi: 10.1016/j.pmn.2018.03.001. Epub 2018 Dec 13. PMID 29776873